CLINICAL TRIAL: NCT00721903
Title: 3D Breast Ultrasound In Predicting Response to Breast Cancer Therapies
Brief Title: Three Dimensional (3D) Ultrasound in Predicting Response to Breast Cancer Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul L. Carson Ph.D, Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2001-0124; UMCC 0005 (Other: Univ. of Michigan Comprehensive Cancer Center); P01CA087634 (NIH)
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancers
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Subjects (Active Comparator): Ultrasound scan
  Interventions: Procedure: Ultrasound Scan
- Cancer (Active Comparator): 120 women diagnosed by biopsy to have breast cancer will have an ultrasound scan
  Interventions: Procedure: Mammography and Ultrasound

INTERVENTIONS:
Procedure: Ultrasound Scan — 10 female volunteers with normal breast who will be studied to refine imaging techniques and for comparison with patients. To the degree possible, the volunteer group will be age-matched to patients with symptoms, initially 30 to 70 years of age.
  Arms: Healthy Subjects
Procedure: Mammography and Ultrasound — To determine how well from ultrasound scans, changes in malignant masses can be measured, and to whether the use of a dye visible by ultrasound will be useful in evaluating different therapies for breast cancer.
  Arms: Cancer

SUMMARY:
The purpose of this study is to determine how well changes can be determined in malignant masses from ultrasound scans.

DETAILED DESCRIPTION:
To evaluate the proportions of correct diagnosis of response to breast Cancer therapies for localized breast cancer by ultrasound. To develop a model based on patient characteristics, physical exam, and radiologic studies which will predict the possibility that a patient has had a complete pathological response to chemotherapy neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer prior to receiving breast cancer therapy.
* Diagnosis of breast cancer must be confirmed by fine needle aspiration or core biopsy.

Exclusion Criteria:

* Poorly controlled diabetes.
* Contralateral mastectomy prior to neoadjuvant chemotherapy.
* Not a surgical candidate.
* No previous axillary lymph node dissection.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2000-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Volume change on spatially registered (aligned) images tracks path. response better than volume change on unregistered images. | 2002-2014
  Self explanatory.

SECONDARY OUTCOMES:
Spatially register pre, intra and post treatment ultrasound image volumes of treated tumor. | 2002-2014
  Visually measure separation between two corresponding points in two ultrasound image volumes after registration to verify registration accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Paul L. Carson, Ph.D., Principal Investigator — University of Michigan; Paul Carson, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States